CLINICAL TRIAL: NCT05880797
Title: Multidimensional and Multimodal Profiling of Oropharyngeal Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-69452; NCI-2023-05592 (Registry Identifier: National Cancer Institute Clinical Trials Reporting Program)
Record Dates: First submitted 2023-05-17; First posted 2023-05-30 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Oropharyngeal Carcinoma; Human Papilloma Virus
MeSH Terms: conditions — Oropharyngeal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The investigators propose to collect blood 30-50cc of blood from Pre-treatment up to 36 month post treatment (+/- 6 months or at the closest visit the patient is being seen for their standard of care visit).
  The investigators also will collect tumor sample (FFPE) or fresh tissue post-excision or surgery and also digitize the de-identified tissue slides (H&E and/or HPV biomarker slides). No extra tissue will be taken at time of procedure, this will only be collected, if and when feasible, after the tumor has been removed post procedure.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to better understand the natural history of oropharyngeal carcinoma (OPC), with or without an association with the human papilloma virus (HPV). For this study, the investigators plan to collect blood from OPC patients prior to treatment and at six subsequent time points.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with oropharyngeal carcinoma or patients with cancer of the unknown primary that is HPV associated, or possibly deemed to be originating from the oropharynx.

Exclusion Criteria:

* Not willing to sign consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with known or suspected oropharyngeal carcinoma. All patients with OPC getting surgery at Stanford are invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Sample collection | prior to start of treatment
  30-50cc of blood
Sample collection | up to 36 months post-op
  30-50cc of blood

SECONDARY OUTCOMES:
tumor sample | Day 1
  tumor sample (FFPE) or fresh tissue post-excision or surgery, this will only be collected, if and when feasible, after the tumor has been removed post procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Holsinger, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States